CLINICAL TRIAL: NCT06359327
Title: Effect of Consumption of Pep19 on Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Proteimax Biotechnology Israel LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Pro00075623
Record Dates: First submitted 2024-03-27; First posted 2024-04-11 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Quality of Life; Obesity; Sleep Quality
Keywords: Peptide; Body weight managment; Sleep
MeSH Terms: conditions — Obesity; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Pep19 2 mg (Active Comparator)
  Interventions: Dietary Supplement: Pep19 2 mg
- Pep19 5 mg (Active Comparator)
  Interventions: Dietary Supplement: Pep19 5 mg

INTERVENTIONS:
Dietary Supplement: Placebo — Subjects will be given an informed consent as per the form submitted to Advarra IRB. 8 randomized subjects will be given placebo for 60 days. Placebo will be formulated as a dietary supplement in veggie capsules with microcrystalline cellulose excipient.
  Arms: placebo
Dietary Supplement: Pep19 2 mg — Subjects will be given an informed consent as per the form submitted to Advarra IRB. 8 randomized subjects will be given 2 mg of Pep19 for 60 days. Placebo will be formulated as a dietary supplement in veggie capsules with microcrystalline cellulose excipient.
  Arms: Pep19 2 mg
Dietary Supplement: Pep19 5 mg — Subjects will be given an informed consent as per the form submitted to Advarra IRB. 8 randomized subjects will be given 5 mg of Pep19 for 60 days. Placebo will be formulated as a dietary supplement in veggie capsules with microcrystalline cellulose excipient.
  Arms: Pep19 5 mg

SUMMARY:
Pep19 is a naturally occurring peptide (protein) that triggers loss of body fat. It has been certified Generally Recognized as Safe (GRAS) at up to 3.8 grams per day and may be included in various foods. Pep19 has no effect on the brain, heart, pancreas or skeletal muscle. It is highly purified, not allergenic or mutagenic, and free of microbes, metals and other contaminants. Preliminary, open-label, uncontrolled studies have shown that Pep19 is well tolerated in rodents, dogs, and humans. This placebo-controlled study will evaluate the effects of two doses of Pep19™ -- 2 mg and 5 mg - on quality of life and sleep quality in obese subjects.

DETAILED DESCRIPTION:
Pep19 is a naturally occurring peptide (protein) that triggers loss of body fat. Obesity is a complex, multifactorial disease that develops from the interaction of genetic, metabolic, social, behavioral, and cultural factors. Numerous studies have demonstrated that obese persons experience significant impairments in quality of life as a result of their obesity, with greater impairments associated with greater degrees of obesity. Weight loss has been shown to improve quality of life in obese persons undergoing a variety of treatments.

Quality of life (QoL) is a concept which aims to capture the well-being. For example, common facets of QoL include personal health (physical, mental, and spiritual), relationships, education status, work environment, social status, wealth, a sense of security and safety, freedom, autonomy in decision-making, social-belonging and their physical surroundings. The World Health Organization explains QoL as a subjective evaluation of one's perception of their reality relative to their goals as observed through the lens of their culture and value system. Therefore, if the individual is feeling that its clothes are fitting better and that he is more motivate to lose weight, it could be considered an improvement of QoL.

In this study we will access QoL in two different ways. Using the S-12 questionnaire to assess physical and mental health, in an indirect way, as this is the view that the subject has of himself. And we will also use biomarkers (weight loss, glucose and insulin levels and so on) to obtain subject-independent data on the physiological changes that could be a reason why the subject is feeling better because of Pep19 supplementation. It has been shown that in obese subjects the improvement of QoL is linked with weight loss, which is directly linked to physical health improvement (weight loss, improvement in plasma biomarkers such as glucose and insulin levels and so on).

Another aspect of this study is the influence of Pep19 on sleep quality in obese subjects. There are a lot of studies suggesting an association between obesity and sleep disturbances. The most well study sleep disturbance associated to obesity is sleep apnea, but the increased visceral adipose tissue might be responsible for the secretion of inflammatory cytokines that could contribute to alter the sleep-wake rhythm, which impairs sleep quality. Animal data showed that Pep19 treatment of rats submitted a sugar supplementation (a model of insulin resistance) decrease visceral adipose tissue. Based on the animal data the investigators would like to study if Pep19 could change the sleep quality and if this change is correlated to the changes on body composition and metabolic parameters.

Pep19 has been certified Generally Recognized as Safe (GRAS) at up to 3.8 grams per day and may be included in various foods. Pep19 has no effect on the brain, heart, pancreas or skeletal muscle. It is highly purified, not allergenic or mutagenic, and free of microbes, metals and other contaminants.

Preliminary, open-label, uncontrolled studies have shown that Pep19 is well tolerated in rodents, beagles, and humans. Each of the beagles and humans received 5mg of Pep19 as an oral supplement in the form of a veggie capsule taken daily for 30 days. Each capsule was composed of the Pep19 plus microcrystalline excipient blended into a veggie capsule with composition as described below. No adverse events were observed. The only surprise was that a few of the humans spontaneously reported improved sleep quality.

This placebo controlled study will evaluate the effects of two doses of Pep19™ -- 2 mg and 5 mg - on two primary endpoints: quality of life and sleep quality. The lower 2 mg dose is being tested because analysis of the human data suggests that a lower normalized dose was associated with fat loss and improved sleep quality. It may be that 2mg has the same effect as 5mg and future use can rely on a 60% lower dose.

Objectives - The purpose of this study is to assess changes in quality of life and sleep quality.

ELIGIBILITY:
Inclusion Criteria:

1. Generally healthy adults between the ages of 40 and 60 years of age, i.e., adults who are community living and able to come to the clinic for qualification and followup appointments
2. BMI between 30 and 35 kg/m2

Exclusion Criteria:

1. Pregnancy, lactation
2. Anti-obesity supplements or medications, e.g. semaglutide

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-05-28 (Actual); Primary Completion 2024-07-28 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Improvement on QoL | 60 days
  The study main endpoint is QoL. The study involves standard assessments, in the study will use the questionnaires SF-12 to assess quality of life.
Improvement on Sleep quality | 60 days
  Related to QoL, the study will use the questionnaires PSQI to assess quality of sleep.

SECONDARY OUTCOMES:
Temperature | 60 days
  The study involves standard assessments, in the study will use a thermometer to assess temperature in Celsius degrees.
Blood pressure | 60 days
  In the study will be used a sphygmomanometer to measure blood pressure in mmHg.
Heart rate | 60 days
  In the study will be used a heart rate measuring device to measure heart rate in beats per secound.
circumference | 60 days
  In the study will be used a measuring tape to measure circumference in centimeters.
blood tests | 60 days
  In the study will be used ELISA assay to measure triglycerides, , ALT, AST, C-reactive protein, glucose, insulin, HgBA1c. All results will be express in mmol/L.
Body fat | 60 days
  In de study will be used DEXA scan to measure the porcentage of fat in each subject.
Body weight | 60 days
  In the study we will use a scale to measure the participants' weight in kg.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Haffizulla, MD, Principal Investigator — Precision Clinical Research
Locations (1):
- Precision Clinical Research, LLC, Sunrise, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reckziegel P, Festuccia WT, Britto LRG, Jang KLL, Romao CM, Heimann JC, Fogaca MV, Rodrigues NS, Silva NR, Guimaraes FS, Eichler RAS, Gupta A, Gomes I, Devi LA, Heimann AS, Ferro ES. A novel peptide that improves metabolic parameters without adverse central nervous system effects. Sci Rep. 2017 Nov 1;7(1):14781. doi: 10.1038/s41598-017-13690-9. PMID 29093454
- [Background] Silverio R, Barth R, Heimann AS, Reckziegel P, Dos Santos GJ, Romero-Zerbo SY, Bermudez-Silva FJ, Rafacho A, Ferro ES. Pep19 Has a Positive Effect on Insulin Sensitivity and Ameliorates Both Hepatic and Adipose Tissue Phenotype of Diet-Induced Obese Mice. Int J Mol Sci. 2022 Apr 7;23(8):4082. doi: 10.3390/ijms23084082. PMID 35456900